CLINICAL TRIAL: NCT02067182
Title: Prevention of Silent Cerebral Thromboembolism by Oral Anticoagulation With Dabigatran After Pulmonary Vein Isolation for Atrial Fibrillation
Acronym: ODIn-AF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Georg Nickenig (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor-Investigator, Georg Nickenig, Prof., University Hospital, Bonn
Organization: University Hospital, Bonn (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MED2-201301; 2013-003492-35 (EudraCT Number)
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Atrial Fibrillation; Cardioembolic Events; Oral Anticoagulation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dabigatran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Anticoagulation with Dabigatran (Experimental): The recommended daily dose of Pradaxa is 300 mg taken as one 150 mg capsule twice daily.
  For the following patients the recommended daily dose of Pradaxa is 220 mg taken as one 110 mg capsule twice daily:
  * Patients aged 75 years or above
  * Cr-Cl 30-50 ml/min
  * Patients who receive concomitant verapamil
  For the following groups, the daily dose of Pradaxa of 300 mg or 220 mg should be selected based on an individual assessment of the thromboembolic risk and the risk of bleeding:
  * Patients with moderate renal impairment
  * Patients with gastritis, esophagitis or gastroesophageal reflux
  * Other patients at increased risk of bleeding
  Interventions: Drug: Dabigatran
- No Oral Anticoagulation (No Intervention)

INTERVENTIONS:
Drug: Dabigatran — * Antral pulmonary vein ablation for patients with AF
  * left atrial fibrosis/electrical scar assessment by electroanatomical mapping
  * followed by 6 months OAC (3 months blanking period + 3 months observation period)
  * in case of AF-recurrence in month 4-6: re- pulmonary vein ablation
  * followed again by 6 months OAC (3 months blanking period + 3 months observation period)
  AF-free patients as assessed by 72h Holter ECG and symptoms wil be random-izedals to the following two interventional arms:
  * Experimental arm (group A): OAC with dabigatran for 12 months
  * Control arm (group B): No OAC (no placebo medication) for 12 months - Cerebral MRI at randomisation and 12 months later
  Arms: Oral Anticoagulation with Dabigatran

SUMMARY:
Oral anticoagulation treatment (OAC) following clinically successful catheter abla-tion of atrial fibrillation (AF) is controversial. Recent guidelines recommended con-tinuation of OAC in all patients with CHA2DS2VASc score ≥2 even if there is no evidence of recurrent AF (Camm JA et al., Eur Heart J 2012). The net clinical ben-efit of OAC after successful ablation in these patients remains to some extent un-clear. As OAC bears the risk of bleeding events, the ODIn-AF study aims to evalu-ate the positive effect of OAC on the incidence of silent cerebral embolic events in patients with a high risk for embolic events, free from AF after successful pulmo-nary vein ablation. ODIn-AF aims to determine that continued administration of dabigatran is superior in the preven-tion of silent cerebral embolism to discontinuation of OAC after 3 months in pa-tients free from symptomatic AF-episodes with a CHA2DS2VASc score ≥2 after the first pulmonary vein ablation for paroxysmal AF.

ELIGIBILITY:
Inclusion criteria:

1. Written informed consent
2. Patients undergoing circumferential antral PV ablation for non-valvular (mitral regurgitation less than moderate- severe insufficiency; no relevant mitral stenosis with a mean pressure gradient >5mmHg) symptomatic, paroxysmal AF or persistent AF (duration < 12 months) with risk factors resulting in a CHA2DS2VASc score ≥2, using a cooled tip RF-, laser- or cryo-balloon-catheter.
3. CHA2DS2VASc score ≥2

Randomization criteria:

1. Sinus rhythm (as assessed by 72h Holter ECG) following the 3 months blanking and 3 months observation period after first or second pulmo-nary vein ablation procedure
2. No clinical evidence of recurrent AF after completing 3 months blanking and 3 months observation period as assessed by symptoms
3. No other relevant contraindication for OAC assessed by randomization MRI of the brain

Exclusion criteria:

1. Severe mental retardation or psychiatrical disorder resulting in incapabil-ity to adequately understand nature, significance, implications and risks of study parcipitation (i.e. bipolar disorders, severe depression, suicidal tendencies, among others) as judged by the local physician, ongoing drug or alcohol addiction (> 8 drinks/week)
2. Pregnancy /breast feeding
3. Severely impaired renal function, GFR < 30 ml/min
4. Impaired liver function (ALT/AST transaminase count 3fold higher than normal values) or liver disease with reduced life expectancy <1 year
5. Valvular AF (moderate- severe mitral insufficiency; relevant mitral steno-sis with a mean pressure gradient >5mmHg)
6. Long standing persistent (>12 months) and permanent AF
7. NSTEMI/STEMI/implantated drug eluting stent with indication for dual antiplatelet therapy within 12 months before enrolment
8. History of complex left atrial ablation procedures. One previous PVI al-lowed.
9. Clinical indication for extended left atrial ablation procedures (CFAE-, rotor-ablation)
10. History or presence of left atrial or ventricular thrombus
11. History of stroke / TIA independent from etiology
12. Acute major bleedings
13. Lesion or condition, if considered a significant risk factor for major bleeding. This may include current or recent gastrointestinal ulceration, presence of malignant neoplasms at high risk of bleeding, recent brain or spinal injury, recent brain, spinal or ophthalmic surgery, recent intracranial haemorrhage, known or suspected oesophageal varices, arteriovenous malformations, vascular aneurysms or major intraspinal or intracerebral vascular abnormalities
14. Need for concomitant anitcoagulation in addition to dabigatran
15. History of previous surgery resulting in contraindication for OAC
16. History of malignoma resulting in contraindication for OAC
17. Mechanical prosthetic heart valve or other indication for permanent OAC
18. Contraindication for MRI (i.e. metal implants unsuitable for MRI, wearing of magnetic or metallic objects that cannot be removed from the body (such as body piercing, implanted electrodes, contraceptive coil), inabil-ity to lie on the back for an extended period of time, uncontrollable claustrophobia, hypersensitivity to noise etc.). Pacemaker and ICD-patients may be included at the discretion of the local investigators/radiologists if MRI is warranted
19. Hypersensitivity against dabigatran or other ingredients of the medical product
20. Concomitant medication with dronedarone, ketoconazole, itraconazole, cyclosporine, tacrolimus or other interacting drugs as specified in the drug information
21. Simultaneous participation in any clinical trial involving administration of an investigational medicinal product within 30 days prior to clinical trial beginning
22. Females of childbearing potential, who are not using or not willing to use medically reliable methods of contraception for the entire study duration (such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices) unless they are surgically sterilized / hysterectomized or there are any other criteria considered sufficiently reliable by the investigator in individual cases
23. Conditions which interfere with the study treatment at the discretion of the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-08; Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Incidence of new micro- and macro-embolic lesions on cerebral MRI incl. flare and diffusion weighted imaging 12 months after randomization compared to baseline MRI (3 months after AF catheter ablation) | 12 months

SECONDARY OUTCOMES:
Location, size and number of new micro- and macro-embolic lesions on cerebral MRI | 12 months
Incidence of clinically evident cardio-embolic events (stroke, TIA, systemic embolism) | 12 months
Severity of neurological deficits assessed by Modified Rankin Scale | 12 months
Incidence of other thrombotic or thrombo-embolic events (myocardial in-farction, deep vein thrombosis, pulmonary embolism) | 12 months
Life-threatening / major / minor bleedings | 12 months
Hemorrhagic cerebral infarction | 12 months
All-cause mortality / Cardiovascular mortality | 12 months
Correlation of cardio-embolic events to method used for PVI (cryo-balloon versus RF) | 12 months
Correlation of cardio-embolic events with arrhythmia recurrence (atrial fi-brillation or atrial flutter post ablationem with ECG documentation or symp-toms) | 12 months
Quality of life questionnaire (AF-specific symptoms, SF36) | 12 months
Neuropsychological questionnaire (RBANS A&B) | 12 months
Assessment of neurocognitive deficits: Minimental Test | 12 months

OTHER OUTCOMES:
Major / minor bleeding events | 12 months
Clinically evident cardio-embolic events | 12 months
Serious Adverse Events | 12 months

CONTACTS AND LOCATIONS:
Locations (19):
- Germany (19):
  - Heart Center Freiburg University Bad Krozingen, Bad Krozingen
  - Heart Center Bad Neustadt-Saale, Bad Neustadt an der Saale
  - Bielefeld Clinical Centre, Bielefeld
  - Dept. of Medicine-Cardiology University Clinic Bonn, Bonn
  - University Hospital Cologne, Cologne
  - University Hospital Gießen, Giessen
  - University Hospital Göttingen, Göttingen
  - Hannover Medical School, Hanover
  - Westpfalz-Clinic GmbH Kaiserslautern, Kaiserslautern
  - Municipal Clinical Center Karlsruhe, Karlsruhe
  - St. Vincentius Hospital, Karlsruhe
  - Heart Center Leipzig, Leipzig
  - Ludwigshafen Hospital, Ludwigshafen
  - Hospital Lüdenscheid, Lüdenscheid
  - University Hospital Mannheim, Mannheim
  - Peter Osypka Heart Center, Munich
  - University Hospital Tübingen, Tübingen
  - Schwarzwald-Baar Hospital Villingen Schwenningen, Villingen-Schwenningen
  - Helios Hospital, Wuppertal

REFERENCES:
- [Derived] Schrickel JW, Linhart M, Bansch D, Thomas D, Nickenig G. Rationale and design of the ODIn-AF Trial: randomized evaluation of the prevention of silent cerebral thromboembolism by oral anticoagulation with dabigatran after pulmonary vein isolation for atrial fibrillation. Clin Res Cardiol. 2016 Feb;105(2):95-105. doi: 10.1007/s00392-015-0933-1. Epub 2015 Oct 29. PMID 26514352